CLINICAL TRIAL: NCT03685331
Title: Harnessing Olaparib, Palbociclib and Endocrine Therapy: A Phase I/II Trial of Olaparib, Palbociclib and Fulvestrant in Patients With BRCA Mutation-associated, Hormone Receptor-positive, Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Metastatic Breast Cancer (HOPE)
Brief Title: HOPE: Olaparib, Palbociclib and Fulvestrant in Patients With BRCA Mutation-associated, HR+, HER2-metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 21118
Record Dates: First submitted 2018-09-18; First posted 2018-09-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer; Advanced Breast Cancer; BRCA2 Mutation; BRCA1 Mutation
Keywords: HER2-negative
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; olaparib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: The phase I component is a dose-escalation study. Dose escalation will follow a 3+3 design. An additional cohort of at least 36 patients (total number of patients in phase I and phase II = 54) will be included on the single-arm, non-randomized phase II portion of this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase I Level 0 (Experimental): (28-day cycle)
  Olaparib 300 mg by mouth twice a day, days 1-28; fulvestrant 500 mg intramuscularly, Day 1 + 500 mg intramuscularly Cycle 0 Day 15; palbociclib 75 mg by mouth daily, days 1-21, beginning at cycle 1
  Interventions: Drug: Palbociclib; Drug: Olaparib; Drug: Fulvestrant
- Phase I Level 1 (Experimental): (28-day cycle)
  Olaparib 300 mg by mouth twice a day, days 1-28; fulvestrant 500 mg intramuscularly, Day 1 + 500 mg intramuscularly Cycle 0 Day 15; palbociclib 100 mg by mouth daily, days 1-21, beginning at cycle 1
  Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-mandated study removal.
  Interventions: Drug: Palbociclib; Drug: Olaparib; Drug: Fulvestrant
- Phase I Level 2 (Experimental): (28-day cycle)
  Olaparib 300 mg by mouth twice a day, days 1-28; fulvestrant 500 mg intramuscularly, Day 1 + 500 mg intramuscularly Cycle 0 Day 15; palbociclib 125 mg by mouth daily, days 1-21, beginning at cycle 1
  Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-mandated study removal.
  Interventions: Drug: Palbociclib; Drug: Olaparib; Drug: Fulvestrant
- Phase II (Experimental): (28-day cycle) Olaparib 300 mg by mouth twice a day, days 1-28; fulvestrant 500 mg intramuscularly once monthly on Day 1 of each cycle + 500 mg intramuscularly on Cycle 1 Day 15; palbociclib dose as per maximum tolerated dose determined during Phase I, by mouth daily, days 1-21
  Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-mandated study removal.
  Interventions: Drug: Palbociclib; Drug: Olaparib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Palbociclib — Combination of palbociclib, olaparib, and fulvestrant.
Drug: Olaparib — Combination of palbociclib, olaparib, and fulvestrant.
Drug: Fulvestrant — Combination of palbociclib, olaparib, and fulvestrant.

SUMMARY:
The main purpose of this research study is to learn whether the investigational combination of olaparib, palbociclib, and fulvestrant is safe in patients with estrogen receptor-positive breast cancer and BRCA1 or BRCA2 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Females/males ≥ age 18
* Germline or somatic deleterious or suspected deleterious mutation in BRCA1 or BRCA2
* Metastatic or locally advanced unresectable breast cancer that is ER and/or PR positive (>1%) and HER2 nonamplified
* Prior treatment with 0-2 prior lines of chemotherapy for metastatic breast cancer
* Regarding prior platinum-based chemotherapy:

  1. Patients who received prior platinum-based chemotherapy in the adjuvant or neoadjuvant setting for breast cancer are eligible if treatment was completed at least 12 months prior to diagnosis of metastatic disease.
  2. Patients who received platinum for advanced breast cancer are eligible to enter the study provided there was no evidence of disease progression during the platinum chemotherapy.
  3. Patients who received prior platinum-based as a potentially curative treatment for a prior non-breast cancer (e.g., ovarian cancer) with no evidence of disease for 5 years or greater prior to study entry are permitted.
* Deemed a candidate for endocrine therapy (any prior endocrine therapy is permitted; no prior endocrine therapy is also permitted)
* Adequate organ and bone marrow function
* ECOG performance status 0-1
* At least one measurable disease or disease that can be assessed by CT or MRI
* Life expectancy ≥ 16 weeks
* Postmenopausal as defined below. Women who are on pharmacologic ovarian suppression must have two negative urine or serum pregnancy tests: one during screening (within 28 days prior to study treatment) and one within 7 days prior to commencing treatment.

Postmenopausal is defined as one of the below:

* Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
* Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
* radiation-induced oophorectomy with last menses >1 year ago
* chemotherapy-induced menopause with >1 year interval since last menses
* bilateral oophorectomy or hysterectomy
* on luteinizing hormone-releasing hormone (LHRH) agonists according to current clinical practice standards as pharmacologic ovarian suppression
* Female patients of childbearing potential (not post-menopausal as defined above) must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 1 month after last dose of study drug(s) to prevent pregnancy.
* Male patients and their sexual partners of childbearing potential must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner.
* Willing to comply with study requirements and procedures including use of appropriate contraception, willingness to discontinue herbal preparations / medications, and study biopsy if archival tissue is not available

Exclusion Criteria:

* Involvement in study planning or conduct
* Regarding prior olaparib or palbociclib,

  a) Phase II: Patients who previously progressed on olaparib or palbociclib for metastatic breast cancer treatment are excluded
* Participation in another clinical study with an investigational product during the last 3 weeks
* Systemic chemotherapy or radiotherapy (except palliative) within 3 weeks of start of study treatment
* Major surgery within 2 weeks of start of study treatment
* Other malignancy within the last 5 years with exceptions listed in the protocol
* Concomitant strong or moderate CYP3A inhibitors/ inducers
* Persistent toxicity of prior cancer therapy that is grade ≥ 2 except for alopecia or neuropathy
* MDS or features suggestive of MDS/AML
* Symptomatic uncontrolled brain metastases
* Patients considered to be at poor medical risk
* QTc >470 msec on 2 or more time points or a family history of long QT syndrome
* Unable to swallow or absorb oral medication
* Immunocompromised patients
* Pregnant or breast-feeding
* Hypersensitivity to olaparib, palbociclib, fulvestrant, or any excipients of these products
* Known active hepatitis
* Prior bone marrow transplant
* Whole blood transfusions 120 days prior to signing consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From first dose of protocol therapy to progression or death due to any cause, whichever comes first, an estimated average of 7 months

SECONDARY OUTCOMES:
Objective response rate | From first dose of protocol therapy to progression or death due to any cause, whichever comes first, an estimated average of 7 months
  Includes complete and partial response as per RECIST 1.1 criteria. Overall response rate will be defined as the proportion of patients within the efficacy analysis set that experience a complete or partial response.
24-week clinical benefit rate | From the date of study treatment until the date of progression, an estimated average of 7 months
  Defined as the proportion of patients within the efficacy analysis set that experience clinical benefit ≥24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Payal D. Shah, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bruno L, Ostinelli A, Waisberg F, Enrico D, Ponce C, Rivero S, Blanco A, Zarba M, Loza M, Fabiano V, Amat M, Pombo MT, Noro L, Chacon M, Colo F, Chacon R, Nadal J, Nervo A, Costanzo V. Cyclin-Dependent Kinase 4/6 Inhibitor Outcomes in Patients With Advanced Breast Cancer Carrying Germline Pathogenic Variants in DNA Repair-Related Genes. JCO Precis Oncol. 2022 Mar;6:e2100140. doi: 10.1200/PO.21.00140. PMID 35235412